CLINICAL TRIAL: NCT03220126
Title: An Assessment of the Absolute and Relative Bioavailability of Subcutaneous Doses of LY3074828 When Coadministered With LY9999QS to Healthy Subjects
Brief Title: A Study to Assess the Amount of LY3074828 That Gets Into the Body When Given With LY9999QS, in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 16861; I9O-MC-AABA (Other: Eli Lilly and Company); 2017-001242-10 (EudraCT Number)
Record Dates: First submitted 2017-07-14; First posted 2017-07-18 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Healthy
MeSH Terms: interventions — mirikizumab

STUDY DESIGN:
Intervention Model Description: Treatments 2 and 3 of LY900021 will be administered in parallel with LY3074828. Treatments 2, 3, and 4 of LY900021 will be administered sequentially pending a safety review after administration of Treatments 2 and 3.
Masking Description: Open
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- LY3074828 - Treatment 1 (Experimental): Single intravenous (IV) dose of LY3074828
  Interventions: Biological: LY3074828
- LY900021 - Treatment 2 (Experimental): Single subcutaneous (SC) dose of LY900021 (LY3074828 coadministered with LY9999QS)
  Interventions: Biological: LY900021
- LY900021 - Treatment 3 (Experimental): Single SC dose of LY900021 (LY3074828 coadministered with LY9999QS)
  Interventions: Biological: LY900021
- LY900021 - Treatment 4 (Experimental): Single SC dose of LY900021 (LY3074828 coadministered with LY9999QS)
  Interventions: Biological: LY900021

INTERVENTIONS:
Biological: LY3074828 — Administered IV
  Arms: LY3074828 - Treatment 1
Biological: LY900021 — Administered SC
  Arms: LY900021 - Treatment 2; LY900021 - Treatment 3; LY900021 - Treatment 4

SUMMARY:
The purpose of this study is to look at the amount of the study drug, LY3074828, that gets into the blood stream and how long it takes the body to get rid of LY3074828 when given together with LY9999QS compared to LY3074828 alone. The tolerability of the different formulations will also be evaluated and information about any side effects experienced will be collected.

Screening is required within 28 days prior to the start of the study. For each participant the total duration of the clinical trial will be approximately 13 weeks, not including screening.

ELIGIBILITY:
Inclusion Criteria:

* Have venous access sufficient to allow for blood sampling and administration of investigational product
* Have clinical laboratory test results within normal reference range for the investigative site, or results with acceptable deviations that are judged to be not clinically significant by the investigator

Exclusion Criteria:

* Must not have an average weekly alcohol intake that exceeds 21 units/week (males) and 14 units/week (females)
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live vaccine(s) (including attenuated live vaccines and those administered intranasally) within 1 month of screening, or intend to during the study
* Must not be immunocompromised
* Must not have known hypersensitivity to hyaluronidases
* Must not have received treatment with biologic agents (e.g. monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Must not have significant allergies to humanised monoclonal antibodies
* Must not have clinically significant multiple or severe drug allergies, or intolerance to topical corticosteroids, or sever post treatment hypersensitivity reactions
* Must not have had lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years
* Must not have had breast cancer within the past 10 years

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area Under the Concentration versus Time Curve (AUC) of LY3074828 | Baseline through Day 85
  PK: AUC of LY3074828

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leeds, United Kingdom